CLINICAL TRIAL: NCT04220203
Title: A Multicenter, Open-label, Treatment Protocol of Tucatinib in Combination With Capecitabine and Trastuzumab in Patients With Previously Treated Unresectable Locally Advanced or Metastatic HER2+ Breast Carcinoma
Brief Title: Treatment Protocol of Tucatinib With Capecitabine and Trastuzumab in Patients With Unresectable Previously Treated HER2+ Breast Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Other Study IDs: SGNTUC-021
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — tucatinib; Capecitabine; Trastuzumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Tucatinib — 300 mg orally two times per day
Drug: Capecitabine — 1000 mg/m^2 orally two times per day on Days 1-14 of each 21-day cycle
Drug: Trastuzumab — Loading dose of 8 mg/kg into the vein (IV; intravenously), followed by 6 mg/kg IV once per 21-day cycle

SUMMARY:
The purpose of this program is to provide access to tucatinib in the United States before FDA approval.

Participants will receive a combination treatment of capecitabine, trastuzumab, and tucatinib. All treatments will be given on a 21 day cycle.

To learn more about this program, contact Seattle Genetics' Medical Information (medinfo@seagen.com).

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed HER2+ breast carcinoma, with HER2+ defined by ISH or FISH or IHC methodology
* For patients WITHOUT presence or history of brain metastases, have received previous treatment with trastuzumab, pertuzumab, and T-DM1
* For patients WITH presence or history of brain metastases, have received previous treatment with trastuzumab
* Have progression of unresectable locally advanced or metastatic breast cancer after last systemic therapy (as confirmed by treating physician), or be intolerant of last systemic therapy
* Have measurable disease or non-measurable disease assessable by standard of care imaging methods
* Have ECOG PS 0 or 1
* Have a life expectancy of at least 6 months, in the opinion of the treating physician

Exclusion Criteria:

* Eligible for a tucatinib clinical trial
* Disease recurrence within 3 months of last capecitabine for metastatic disease
* History of allergic reactions to trastuzumab, capecitabine, or compounds chemically or biologically similar to tucatinib, except for Grade 1 or 2 infusion related reactions to trastuzumab that were successfully managed, or known allergy to one of the excipients in the protocol drugs
* Have received treatment with any systemic anti-cancer therapy (excluding hormonal therapy), non-CNS radiation, or experimental agent ≤ 3 weeks of first dose of protocol treatment or are currently participating in an interventional clinical trial. Have received hormonal therapies <1 week of the first dose of protocol treatment.
* Have any toxicity related to prior cancer therapies that has not resolved to ≤ Grade 1, with the following exceptions:

  * Alopecia and neuropathy, which must have resolved to ≤ Grade 2
  * CHF, which must have been ≤ Grade 1 in severity at the time of occurrence, and must have resolved completely
  * Anemia, which must have resolved to ≤ Grade 2
* Have clinically significant cardiopulmonary disease
* Have known myocardial infarction or unstable angina within 6 months prior to first dose of protocol treatment
* Are known carriers of Hepatitis B or Hepatitis C or have other known chronic liver disease with uncontrolled disease
* Are known to be positive for HIV with uncontrolled disease
* Are pregnant, breastfeeding, or planning a pregnancy
* Require therapy with warfarin or other coumarin derivatives (non-coumarin anticoagulants are allowed)
* Have inability to swallow pills or significant gastrointestinal disease which would preclude the adequate oral absorption of medications
* Have used strong CYP2C8 inhibitor within 5 half-lives of the inhibitor, or have used a CYP2C8 or CYP3A4 inducer within 5 day prior to start of tucatinib treatment.
* Have known dihydropyrimidine dehydrogenase deficiency
* Have evidence within 2 years of the start of protocol treatment of another malignancy that required systemic treatment.

CNS Exclusion - patients must not have any of the following:

* Any untreated brain lesions > 2.0 cm in size, unless discussed with medical monitor and approval for enrollment is given
* Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent). However, patients on a chronic stable dose of ≤ 2 mg total daily of dexamethasone (or equivalent) may be eligible with discussion and approval by the medical monitor
* Any brain lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where increase in size or possible treatment-related edema may pose risk to patient (e.g. brain stem lesions).
* Known or suspected LMD as documented by the treating physician
* Have poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to brain metastases notwithstanding CNS-directed therapy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult